CLINICAL TRIAL: NCT05844150
Title: A Phase II Clinical Trial to Evaluate the Efficacy and Safety of PM8002 in Combination With Etoposide and Platinum in First-line Treatment of Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of PM8002 (Anti-PD-L1/VEGF) in Combination With Chemotherapy in Patients With ES-SCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM8002-BC011C-SCLC-R
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: SCLC
Keywords: ES-SCLC
MeSH Terms: interventions — Platinum; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM8002+Etoposide＋platinum (Experimental): Subjects will be administered with PM8002 plus Etoposide and platinum via intravenously (IV) Q3W for 4 cycles, followed by PM8002 until progression or for a maximum of 2 years.
  Interventions: Drug: PM8002; Drug: Platinum; Drug: Etoposide

INTERVENTIONS:
Drug: PM8002 — IV infusion
Drug: Platinum — IV infusion
Drug: Etoposide — IV infusion

SUMMARY:
PM8002 is a bispecific antibody targeting PD-L1 and VEGF. This study to evaluate the efficacy and safety of PM8002 in combination with etoposide and platinum in first-line treatment of extensive-stage small cell lung cancer

DETAILED DESCRIPTION:
The study is divided into two parts.

The first part is single-arm study, 50 participants were enrolled as of 21 Nov 2023，and recruitment was completed.

The second part is randomized, double-blind study, active controlled design , which will be integrated to another global III study （NCT06712355）.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form before any trial-related processes;
2. Age ≥18 years;
3. Histologically or cytologically confirmed ES-SCLC;
4. No prior systemic therapy for ES-SCLC;
5. Have adequate organ function;
6. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1;
7. Life expectancy of ≥12 weeks;
8. Had at least one measurable tumor lesion according to RECIST v1.1.

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed SCLC;
2. History of severe allergic disease, severe drug allergy or have known allergy to any component of the study drugs;
3. The toxicity of previous anti-tumor therapy has not been alleviated；
4. Have received anti-platelet therapy within 10 days prior to the first dose of the study drugs;
5. Evidence and history of severe bleeding tendency;
6. History of severe cardiovascular diseases within 6 months;
7. Current presence of uncontrolled pleural, pericardial, and peritoneal effusions;
8. History of allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation;
9. History of alcohol abuse, psychotropic substance abuse or drug abuse;
10. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome;
11. Pregnant or lactating women;
12. Other conditions considered unsuitable for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.
Progression free survival (PFS) | Up to approximately 2 years
  Progression free survival (PFS) is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease (SD) based on RECIST v1.1.
Duration of response (DOR) | Up to approximately 2 years
  DOR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Time to response (TTR) | Up to approximately 2 years
  TTR is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieve CR or PR (based on RECIST v1.1).
Pharmacokinetic (PK) parameters | Up to 30 days after last treatment
  The PK parameters including serum concentrations of PM8002 at different time points after study drug administration.
Anti-drug antibody (ADA) | Up to 30 days after last treatment
  To evaluate the incidence of ADA to PM8002.
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (17):
- China (17):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Hospital, Hefei
  - Central Hospital Affiliated To Shandong First Medical University, Jinan
  - Hebei Petro China Central Hospital, Langfang
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Shandong Cancer Hospital, Shandong
  - Shanghai Pulmonary Hospital, Shanghai
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract,articles or papers) or any presentations
Time Frame: After the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.